CLINICAL TRIAL: NCT03203655
Title: Efficacy of a Culturally Sensitive and Linguistically Appropriate Internet and Mobile-based Weight Loss Therapy in Obese Hispanic/Latino Adult Women
Brief Title: Text Based Mobile Technology and Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201704048
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Obesity
Keywords: Mobile text; Obesity; Hispanic; Women
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will be enrolled in the CareMessage™ Adult Obesity texting program, which sends a text message 3 to 5 times a week, encouraging lifestyle modifications (diet and exercise education, and behavioral strategies) that can lead to healthy weight loss.
  Interventions: Behavioral: CareMessage™
- Control Group (Other): The control group will receive the control condition. They will hear an initial talk about weight loss but will not be enrolled in any program or intervention.
  Interventions: Behavioral: Control Condition

INTERVENTIONS:
Behavioral: CareMessage™ — Adult Obesity texting program, which sends a text message 3 to 5 times a week, encouraging lifestyle modifications (diet and exercise education, and behavioral strategies) that can lead to healthy weight loss.
  Arms: Intervention Group
Behavioral: Control Condition — Control condition will receive an initial talk about weight loss but will not be enrolled in any program or intervention.
  Arms: Control Group

SUMMARY:
Hispanic populations in the US are dis-proportionally affected by high rates of obesity and diabetes; according to the Centers for Disease Control and Prevention, Latinos are the minority group with the second-highest obesity prevalence in adults. In comparison to the general female population (61.2%), Mexican American women (73%) have a greater overweight or obese percentage. In addition, more than 50% of Hispanic men and women are expected to develop type-2 diabetes over their lifetime, compared to 40% among whites. Hispanics are also 50% more likely to die from diabetes compared to whites. In many cases Hispanic populations do not have the knowledge, self-confidence and resources to participate in mainstream physical activity and nutrition interventions, which are usually geared towards the general population without considering cultural and linguistic differences.

Information and communication technologies in the form of Internet and mobile phone access have grown enormously during the past decade; these technologies have the potential to affect food intake and physical activity as well as weight loss. Approximately 95% of countries have mobile telephone networks and about 70% of people worldwide use mobile phones.

CareMessage is a Google-backed 501(c)3 nonprofit technology organization based in San Francisco that uses 'smart' text and voice messaging to enable clinical staff to provide automated yet personalized support to patients struggling with chronic conditions. The CareMessage™ Adult Obesity texting program adapts the Health Belief Model by strategically implementing behavioral concepts to help improve self-efficacy.

The investigators will pilot test its effectiveness among a sample of Hispanic women who are at risk of obesity and diabetes by sending a culturally-sensitive and linguistically-appropriate text-based message three to 5 times a week, encouraging lifestyle modifications (diet and exercise education and behavior modification).

DETAILED DESCRIPTION:
The investigators will collect data on 40 obese (Body Mass Index 30-45) Hispanic women ages 21 to 65 years. The purpose of this research study is to test the efficacy of a mobile phone text message-based intervention on weight loss.

After verifying eligibility and enrolling in the study, participants will come to Washington University School of Medicine, at Barnes-Jewish Hospital and fill out some questionnaires. The investigators will perform a brief exam that measures the lean and fat tissue using Dual Energy x-ray Absorptiometry (DXA) technology and will also do a modified 3-hour oral glucose tolerance test (MOGTT).

Participants will wear an accelerometer (activity monitor) over a 7-day period at the beginning (before being randomized and enrolled in the intervention) and at the end of the study.

Half of the participants will be randomized to the intervention group. The intervention group will be enrolled in the CareMessage™ Adult Obesity texting program, which sends a text message 3 to 5 times a week, encouraging lifestyle modifications (diet and exercise education, and behavioral strategies) that can lead to healthy weight loss. The control group will receive an initial talk about weight loss but will not be enrolled in any program or intervention.

After six months have passed, participants will return to Washington University School of Medicine, regardless of the group they were assigned to, for two final visits (a short one, to pick up another activity monitor seven days before the study ends, and a longer visit, to do some final testing and fill out some questionnaires).

ELIGIBILITY:
Inclusion Criteria (for both control and intervention groups)

* Women between 18 21 and 65 years old,
* Poor to normal English literacy,
* Of Hispanic or Latin American origin,
* Having access to a smart phone,
* Obese (BMI 30-45).
* Non-institutionalized population,
* Currently not involved in any other weight loss program,
* Sedentary population (exercising less than 90 minutes per week).

For the phone screening we will need the following data elements:

* Female
* BMI
* Age
* Ethnicity

Exclusion Criteria (for both groups):

* Participants with a history of and/or current mental or physical disabilities.
* Participants with BMI over 45

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Body mass Index | 6 months
  is a measure of body fat based on height and weight that applies to adult men and women.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Parra, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No